CLINICAL TRIAL: NCT02760329
Title: A NOVEL Observational longiTudinal studY on Patients With Asthma and/or COPD to Describe Patient Characteristics, Treatment Patterns and the Burden of Illness Over Time and to Identify Phenotypes and Endotypes.
Brief Title: Observational Study of Obstructive Lung Disease (NOVELTY)
Acronym: NOVELTY
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Other Study IDs: D2287R00103
Record Dates: First submitted 2016-04-05; First posted 2016-05-03 (Estimated); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Asthma; COPD; Chronic Obstructive Pulmonary Disease
Keywords: asthma; COPD; chronic obstructive pulmonary disease; lung disease; chronic airways disease; obstructive lung disease
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Lung Diseases; Lung Diseases, Obstructive | interventions — Blood Specimen Collection; Urination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biomarkers from blood samples including assessment of haematology and collection for storage of serum, plasma, deoxyribonucleic acid (DNA), ribonucleic acid (RNA) and urine samples. Collection of blood and urine samples is optional and will be covered in a separate section of the informed consent form.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic airways disease: Patients with suspected or primary diagnosis of asthma or COPD
  Interventions: Procedure: Blood draw; Procedure: Urine; Procedure: Lung function measurements; Procedure: Fractional Exhaled Nitric Oxide (FENO)

INTERVENTIONS:
Procedure: Blood draw — Biomarkers analyses
Procedure: Urine — Biomarker analyses
Procedure: Lung function measurements — FEV1, FVC, PEF, FEF25-75%, IC, calculated FEV1/FVC ratio and calculated FEV1 % predicted
Procedure: Fractional Exhaled Nitric Oxide (FENO) — Measures level of exhaled nitric oxide.

SUMMARY:
The NOVEL Observational longiTudinal studY (NOVELTY) is an observational study of obstructive lung disease and is a multi-country, multi-centre, prospective, longitudinal cohort study which will recruit patients with a diagnosis, or suspected diagnosis, of asthma and/or Chronic Obstructive Pulmonary Disease (COPD). Patients will undergo clinical assessments and receive standard medical care as determined by their treating physician. Patients enrolled in NOVELTY will be followed up yearly by their treating physician for a total duration of three years. In addition, patients will be followed up remotely every 3 months. The NOVELTY study will collect data currently lacking to allow for multinational data collection to fill regional/local gaps and improve comparability across regions.

DETAILED DESCRIPTION:
The NOVELTY study is a multi-country, multicentre, observational, prospective, longitudinal cohort study which will include patients with a physician diagnosis, or suspected diagnosis, of asthma and/or COPD. Patients will undergo clinical assessments and receive standard medical care as determined by the treating physician. All patients enrolled in the NOVELTY study will be followed up yearly by their treating physician for a total duration of three years. In addition, patients are expected to be followed up remotely once every quarter.

It is estimated that approximately 7,700 patients with suspected or primary diagnosis of asthma and 7,100 patients with suspected or primary diagnosis of COPD will be enrolled by a diverse set of physicians (e.g. primary care physicians, allergists, pulmonologists) from community and hospital outpatient settings within the countries targeted for NOVELTY.

Exposure(s):

The NOVELTY study is a longitudinal cohort study which does not involve or study a specific medicinal product; it will constitute a disease registry. Information about exposure to treatments as part of routine care will be collected (frequency, treatment, duration).

Sample Size Estimations:

The target minimum number of 100 patients per diagnostic label (asthma or COPD), physician-assessed severity level and country has been chosen to support many basic local reimbursement specific requirements with reasonable precision, and to provide large sample size for scientific questions applicable across severities and countries. Therefore, considering the targeted countries, it is estimated that approximately 7,700 patients with asthma and 7,100 patients with COPD will be enrolled.

Statistical Analysis:

After baseline data collection and each annual data collection, data will be summarized for the population overall and by pre specified subgroups, including by country, demographics, exposures, symptom history, treatment history, concurrent clinical features, treatment setting, socioeconomic setting and access to healthcare, where relevant.

Patients' changes regarding their treatment, disease or severity among and other variables that are observed between baseline and follow-up visits, will also be described.

To identify potential differences in disease diagnosis and severity classifications between physicians and guidelines, data collected on lung function results, symptom questionnaires, exacerbation occurrences and medication will allow the formal and consistent classification of the patients according to relevant international guidelines and other current and future phenotypic/diagnostic classifications.

Multivariable models will be used to assess the following: the occurrence of exacerbations and other conditions, including upper and lower Respiratory Tract Infections (RTIs) and their relationship with clinical outcomes, the relationship between Patient Reported Outcomes (PRO) and disease control with impact on daily activity and quality of life, and the relationship between healthcare resource use overall and related to respiratory diseases with disease severity, clinical outcomes, disease type, etc.

Multivariable analysis techniques will be used to identify phenotypes and endotypes, based on biomarkers and/or clinical parameters that are associated with differential outcomes for symptom burden, clinical evolution and healthcare utilisation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis, or suspected diagnosis, of asthma and/or COPD, according to clinician's judgment
* Age: 12 years or older (note: in most countries it will only be feasible to include patients aged 18 years or older)
* Willing and able to sign written, informed consent (or having a responsible, legally authorised representative acting on patient's behalf)
* Enrolment from an active clinical practice

Exclusion Criteria:

* Patients who participated in any respiratory interventional trial during the 12 months prior to enrolment or at enrolment
* Patients who, in the opinion of the physician, are unlikely to complete 3 years of follow-up, e.g. poor literacy, substance abuse, life-threatening co-morbidity
* Patients whose primary respiratory diagnosis (i.e. the condition causing most of their respiratory symptoms) is not asthma or COPD (however, a co-diagnosis of another respiratory disease such as bronchiectasis or interstitial lung disease together with asthma or COPD will be accepted)

In addition, the following are considered criteria for exclusion from the exploratory genetic research (donation of blood for DNA and RNA analysis)

* Previous allogeneic bone marrow transplant
* Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection

Ages: 12 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with suspected or primary diagnosis of asthma and with suspected or primary diagnosis of COPD will be enrolled by a diverse set of physicians (e.g. primary care physicians, allergists, pulmonologists) from community and hospital outpatient settings.
Sampling Method: Probability Sample
Enrollment: 12255 (Actual)
Dates: Start 2016-07-25 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Spirometry - change in Forced Expiratory Volume in 1 second (FEV1) (Litres [L]) | Change from baseline FEV1 at Year 1, 2 and 3
  Lung function test
Spirometry - change in Forced Vital Capacity (FVC) (L) | Change from baseline FVC at Year 1, 2 and 3
  Lung function test
Spirometry - change in Peak Expiratory Flow (PEF) (Litre/second [L/s]) | Change from baseline PEF at Year 1, 2 and 3
  Lung function test
Spirometry - change in Forced Expiratory Flow at 25-75% of the forced vital capacity (FEF25-75%) (L/s) | Change from baseline FEF25-75% at Year 1, 2 and 3
  Lung function test
Spirometry - change in Inspiratory Capacity (IC) (L) | Change from baseline IC at Year 1, 2 and 3
  Lung function test
Post-bronchodilator spirometry - FEV1 (L) | Baseline
  Bronchodilator reversibility test
Post-bronchodilator spirometry - FVC (L) | Baseline
  Bronchodilator reversibility test
Post-bronchodilator spirometry - PEF (L/s) | Baseline
  Bronchodilator reversibility test
Post-bronchodilator spirometry - FEF25-75% (L/s) | Baseline
  Bronchodilator reversibility test
Post-bronchodilator spirometry - IC (L) | Baseline
  Bronchodilator reversibility test
Fractional exhaled nitric oxide (FeNO) (parts per billion [ppb]) | Baseline
  Test to measure fractional exhaled nitric oxide (ppb) levels in exhaled breath
Change in symptoms/symptom control assessed by the Chronic Airways Assessment Test (CAAT) | Change from baseline CAAT scores at Year 1, 2, and 3
  Patient reported outcome questionnaire
Symptoms/symptom control assessed by the modified Medical Research Council (mMRC) scale | Baseline
  Patient reported outcome questionnaire
Change in symptoms/symptom control assessed by the Respiratory Symptoms Questionnaire (RSQ) | Change from baseline RSQ scores at Year 1, 2 and 3
  Patient reported outcome questionnaire
Change in symptoms/symptom control assessed by the Asthma Control Test (ACT) | Change from baseline ACT scores at Year 1, 2 and 3
  Patient reported outcome questionnaire
COPD Foundation Primary Care Tool for Undiagnosed Respiratory Disease and Exacerbation Risk (CAPTURE) - to identify undiagnosed patients with clinically significant COPD | Baseline
  Patient reported outcome questionnaire

CONTACTS AND LOCATIONS:
Locations (288):
- United States (36):
  - Research Site, Loma Linda, California
  - Research Site, Long Beach, California
  - Research Site, Roseville, California
  - Research Site, Aurora, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Clearwater, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Miami, Florida
  - Research Site, Plantation, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Normal, Illinois
  - Research Site, Hutchinson, Kansas
  - Research Site, Shreveport, Louisiana
  - Research Site, Fall River, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Buckley, Michigan
  - Research Site, Hamtramck, Michigan
  - Research Site, Lincoln, Nebraska
  - Research Site, Highland Park, New Jersey
  - Research Site, West Berlin, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, New York, New York
  - Research Site, Rockville Centre, New York
  - Research Site, The Bronx, New York
  - Research Site, Fargo, North Dakota
  - Research Site, Cincinnati, Ohio
  - Research Site, Kettering, Ohio
  - Research Site, Wooster, Ohio
  - Research Site, Altoona, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Austin, Texas
  - Research Site, Houston, Texas
  - Research Site, Live Oak, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Charleston, West Virginia
- Argentina (10):
  - Research Site, Monte Grande, Buenos Aires
  - Research Site, Pilar, Buenos Aires
  - Research Site, Tandil, Buenos Aires
  - Research Site, Buenos Aires, Buenos Aires F.D.
  - Research Site, Concepción del Uruguay, Entre Ríos Province
  - Research Site, San Salvador, Entre Ríos Province
  - Research Site, San Miguel de Tucumán, Tucumán Province
  - Research Site, Buenos Aires
  - Research Site, Córdoba
  - Research Site, Mendoza
- Australia (22):
  - Research Site, Blacktown, New South Wales
  - Research Site, Camperdown, New South Wales
  - Research Site, Coffs Harbour, New South Wales
  - Research Site, Concord, New South Wales
  - Research Site, Kanwal, New South Wales
  - Research Site, Kingswood, New South Wales
  - Research Site, Liverpool, New South Wales
  - Research Site, Miranda, New South Wales
  - Research Site, New Lambton, New South Wales
  - Research Site, Randwick, New South Wales
  - Research Site, Sedney, New South Wales
  - Research Site, Wamberal, New South Wales
  - Research Site, Brisbane, Queensland
  - Research Site, Redcliffe, Queensland
  - Research Site, South Brisbane, Queensland
  - Research Site, Bedford Park, South Australia
  - Research Site, Happy Valley, South Australia
  - Research Site, Woodville South, South Australia
  - Research Site, Frankston, Victoria
  - Research Site, Parkville, Victoria
  - Research Site, Crawley, Western Australia
  - Research Site, Spearwood, Western Australia
- Brazil (5):
  - Research Site, Goiânia, Goiás
  - Research Site, Uberlândia, Minas Gerais
  - Research Site, Blumenau, Santa Catarina
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Canada (13):
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, New Brunswick, New Brunswick
  - Research Site, Burlington, Ontario
  - Research Site, Downsview, Ontario
  - Research Site, Fort Erie, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Québec
- China (23):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Sichuan, Chengdu
  - Research Site, Dongguan, Guangdong
  - Research Site, Shantou, Guangdong
  - Research Site, Shenzhen, Guangdong
  - Research Site, Guangdong, Guangzhou
  - Research Site, Changshacun, Henan
  - Research Site, Zhengzhou, Henan
  - Research Site, Shiyan, Hubei
  - Research Site, Baotou, Inner Mongolia
  - Research Site, Hohhot, Inner Mongolia
  - Research Site, Nanjing, Jiangsu
  - Research Site, Suzhou, Jiangsu
  - Research Site, Yangzhou, Jiangsu
  - Research Site, Nanchang, Jiangxi
  - Research Site, Changchun, Jilin
  - Research Site, Yanji, Jilin
  - Research Site, Xi'an, Shaanxi
  - Research Site, Jinan, Shandong
  - Research Site, Weifang, Shandong
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Hangzhou, Zhejiang
  - Research Site, Jinhua, Zhejiang
- Colombia (6):
  - Research Site, Bogotá, Bogota D.C.
  - Research Site, Bucaramanga, Bogota D.C.
  - Research Site, Manizales, Caldas Department
  - Research Site, Zipaquirá, Cundinamarca
  - Research Site, Villavicencio, Meta Department
  - Research Site, Antioquia
- Denmark (2):
  - Research Site, Aarhus N, Central Jutland
  - Research Site, Viby J, Central Jutland
- France (26):
  - Research Site, Pau, Aquitaine
  - Research Site, Lyon, Auvergne-Rhône-Alpes
  - Research Site, Clermont-Ferrand, Auvergne
  - Research Site, Strasbourg, Bas-Rhin
  - Research Site, Brest, Brittany Region
  - Research Site, Caen, Calvados
  - Research Site, Dijon, Côte-d'Or
  - Research Site, Besançon, Franche-Comté
  - Research Site, Pessac, Gironde
  - Research Site, Mulhouse, Haut-Rhin
  - Research Site, Limoges, Haute-Vienne
  - Research Site, Tarbes, Hautes-Pyrénées
  - Research Site, Montpellier, Hérault
  - Research Site, Orléans, Loiret
  - Research Site, Nancy, Meurthe-et-Moselle
  - Research Site, Bersée, Nord
  - Research Site, Lille, Nord
  - Research Site, Aix-en-Provence, Provence-Alpes-Côte d'Azur Region
  - Research Site, Biarritz, Pyrénées-Atlantiques
  - Research Site, Villefranche-sur-Saône, Rhône
  - Research Site, Le Mans, Sarthe
  - Research Site, Montvilliers, Seine-Maritime
  - Research Site, Rouen, Seine-Maritime
  - Research Site, Créteil, Val-de-Marne
  - Research Site, Paris
  - Research Site, Paris, Île-de-France Region
- Germany (17):
  - Research Site, Bruchsal, Baden-Wurttemberg
  - Research Site, Heidelberg, Baden-Wurttemberg
  - Research Site, Augsburg, Bavaria
  - Research Site, Munich, Bavaria
  - Research Site, Marburg, Hesse
  - Research Site, Peine, Lower Saxony
  - Research Site, Ibbenbueren, North Rhine-Westphalia
  - Research Site, Ratingen, North Rhine-Westphalia
  - Research Site, Dillingen, Saarland
  - Research Site, Dresden, Saxony
  - Research Site, Leipzig, Saxony
  - Research Site, Halberstadt, Saxony-Anhalt
  - Research Site, Lübeck, Schleswig-Holstein
  - Research Site, Reinfeld, Schleswig-Holstein
  - Research Site, Schleswig, Schleswig-Holstein
  - Research Site, Berlin
  - Research Site, Hamburg
- Italy (22):
  - Research Site, Chieti, Abruzzo
  - Research Site, Rome, Lazio
  - Research Site, Mantova, Lombardy
  - Research Site, Monza, Milano
  - Research Site, Montescano, Pavia
  - Research Site, Orbassano, Piedmont
  - Research Site, Torre Del Greco (Napoli), Salerno
  - Research Site, Sassari, Sardinia
  - Research Site, Gravina di Catania, Sicily
  - Research Site, Torrette Di Ancona, The Marches
  - Research Site, Catania
  - Research Site, Ferrara
  - Research Site, Florence
  - Research Site, Foggia
  - Research Site, Genova
  - Research Site, Livorno
  - Research Site, Messina
  - Research Site, Modena
  - Research Site, Napoli
  - Research Site, Palermo
  - Research Site, Pordenone
  - Research Site, Roma
- Japan (23):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Kitakyushu, Fukuoka
  - Research Site, Kurume, Fukuoka
  - Research Site, Omuta, Fukuoka
  - Research Site, Itami, Hyōgo
  - Research Site, Kobe, Hyōgo
  - Research Site, Higashiibaraki-gun, Ibaraki
  - Research Site, Kanazawa, Ishikawa-ken
  - Research Site, Yokohama, Kanagawa
  - Research Site, Ishinomaki, Miyagi
  - Research Site, Kishiwada, Osaka
  - Research Site, Matsue, Shimane
  - Research Site, Shizuoka, Shizuoka, Shizuoka
  - Research Site, Shimotsuga-gun, Tochigi
  - Research Site, Chuo-ku, Tokyo
  - Research Site, Kiyose, Tokyo
  - Research Site, Nakano-ku, Tokyo
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Shizuoka
  - Research Site, Toyama
  - Research Site, Yamagata
- Mexico (6):
  - Research Site, Pachuca, Hidalgo
  - Research Site, Guadalajara, Jalisco
  - Research Site, Mexico City, Mexico City
  - Research Site, Monterrey, Nuevo León
  - Research Site, Villahermosa, Tabasco
  - Research Site, México
- Netherlands (11):
  - Research Site, Arnhem, Gelderland
  - Research Site, Nijmegen, Gelderland
  - Research Site, Zutphen, Gelderland
  - Research Site, Horn, Limburg
  - Research Site, Breda, North Brabant
  - Research Site, Veldhoven, North Brabant
  - Research Site, Alkmaar, North Holland
  - Research Site, Enschede, Overijssel
  - Research Site, Rotterdam, South Holland
  - Research Site, Nieuwegein, Utrecht
  - Research Site, Groningen
- Norway (6):
  - Research Site, Jassheim, Akershus
  - Research Site, Lørenskog, Akershus
  - Research Site, Trollåsen, Akershus
  - Research Site, Tananger, Rogaland
  - Research Site, Oslo
  - Research Site, Trondheim
- South Korea (10):
  - Research Site, Daegu, Daegu Gwang'yeogsi
  - Research Site, Chuncheon, Gang'weondo
  - Research Site, Gwangju, Gwangju Gwang'yeogsi
  - Research Site, Anyang-si, Gyeonggido
  - Research Site, Gyeonggi-do, Gyeonggido
  - Research Site, Seongnam-si, Gyeonggido
  - Research Site, Suwon, Gyeonggido
  - Research Site, Incheon, Incheon Gwang'yeogsi
  - Research Site, Jeonju, Jeonrabugdo
  - Research Site, Seoul, Seoul Teugbyeolsi
- Spain (25):
  - Research Site, Palma de Mallorca, Balearic Islands
  - Research Site, Badalona, Barcelona
  - Research Site, Centelles, Barcelona
  - Research Site, Santa Cruz de Tenerife, Canary Islands
  - Research Site, Alcázar de San Juan, Ciudad Real
  - Research Site, Palmones, Cádiz
  - Research Site, Alcalá de Henares, Madrid
  - Research Site, Móstoles, Madrid
  - Research Site, Pozuelo de Alarcón, Madrid
  - Research Site, Torrelaguna, Madrid
  - Research Site, Cartagena, Murcia
  - Research Site, Pamplona, Navarre
  - Research Site, Vigo, Pontevedra
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, Barakaldo, Vizcaya
  - Research Site, Badajoz
  - Research Site, Barcelona
  - Research Site, Burgos
  - Research Site, Granada
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Murcia
  - Research Site, Valladolid
  - Research Site, Zaragoza
- Sweden (5):
  - Research Site, Värnamo, Jönköping County
  - Research Site, Lund, Skåne County
  - Research Site, Stockholm, Stockholm County
  - Research Site, Uppsala, Uppsala County
  - Research Site, Gothenburg, Västra Götaland County
- United Kingdom (20):
  - Research Site, Swansea, Carmarthenshire
  - Research Site, Chelmsford, Essex
  - Research Site, Southampton, Hampshire
  - Research Site, Watford, Hertfordshire
  - Research Site, Middlesbrough, Kensington and Chelsea
  - Research Site, Hull, Kingston Upon Hull, City of
  - Research Site, Thornton-Cleveleys, Lancashire
  - Research Site, London, London, City of
  - Research Site, Wishaw, North Lanarkshire
  - Research Site, York, North Yorkshire
  - Research Site, Belfast, Northern Ireland
  - Research Site, Nottingham, Nottinghamshire
  - Research Site, Tyne and Wear, South Tyneside
  - Research Site, Warwickshire, Warwickshire
  - Research Site, Pickering, York
  - Research Site, Birmingham
  - Research Site, Liverpool
  - Research Site, Manchester
  - Research Site, Newport
  - Research Site, York

REFERENCES:
- [Derived] Papi A, Hughes R, Del Olmo R, Agusti A, Chipps BE, Make B, Tomaszewski E, Peres Da Costa K, Srivastava D, Vestbo J, Janson C, Burgel PR, Price D. Relationships between symptoms and lung function in asthma and/or chronic obstructive pulmonary disease in a real-life setting: the NOVEL observational longiTudinal studY. Ther Adv Respir Dis. 2024 Jan-Dec;18:17534666241254212. doi: 10.1177/17534666241254212. PMID 38841799
- [Derived] Agusti A, Hughes R, Rapsomaki E, Make B, Del Olmo R, Papi A, Price D, Benton L, Franzen S, Vestbo J, Mullerova H. The many faces of COPD in real life: a longitudinal analysis of the NOVELTY cohort. ERJ Open Res. 2024 Feb 12;10(1):00895-2023. doi: 10.1183/23120541.00895-2023. eCollection 2024 Jan. PMID 38348246
- [Derived] Ding B, Chen S, Rapsomaniki E, Quinton A, Cook W, Reddel HK, Papi A; NOVELTY Scientific Community; NOVELTY study investigators. Burden of Uncontrolled Severe Asthma With and Without Elevated Type-2 Inflammatory Biomarkers. J Allergy Clin Immunol Pract. 2024 Apr;12(4):970-982. doi: 10.1016/j.jaip.2023.12.021. Epub 2023 Dec 22. PMID 38141721
- [Derived] Ding B, Chen S, Srivastava D, Quinton A, Cook W, Papi A, Reddel HK; NOVELTY Scientific Community; NOVELTY study investigators. Symptom Burden, Health Status, and Productivity in Patients with Uncontrolled and Controlled Severe Asthma in NOVELTY. J Asthma Allergy. 2023 Jun 11;16:611-624. doi: 10.2147/JAA.S401445. eCollection 2023. PMID 37334017
- [Derived] Hughes R, Rapsomaniki E, Bansal AT, Vestbo J, Price D, Agusti A, Beasley R, Fageras M, Alacqua M, Papi A, Mullerova H, Reddel HK; NOVELTY Scientific Community; NOVELTY study investigators. Cluster Analyses From the Real-World NOVELTY Study: Six Clusters Across the Asthma-COPD Spectrum. J Allergy Clin Immunol Pract. 2023 Sep;11(9):2803-2811. doi: 10.1016/j.jaip.2023.05.013. Epub 2023 May 23. PMID 37230383
- [Derived] Tomaszewski EL, Atkinson MJ, Janson C, Karlsson N, Make B, Price D, Reddel HK, Vogelmeier CF, Mullerova H, Jones PW; NOVELTY Scientific Community; NOVELTY study investigators. Chronic Airways Assessment Test: psychometric properties in patients with asthma and/or COPD. Respir Res. 2023 Apr 8;24(1):106. doi: 10.1186/s12931-023-02394-6. PMID 37031164
- [Derived] Marshall H, Wild JM, Smith LJ, Hardaker L, Fihn-Wikander T, Mullerova H, Hughes R. Functional imaging in asthma and COPD: design of the NOVELTY ADPro substudy. ERJ Open Res. 2023 Apr 3;9(2):00344-2022. doi: 10.1183/23120541.00344-2022. eCollection 2023 Mar. PMID 37020837
- [Derived] Hughes R, Rapsomaniki E, Janson C, Keen C, Make BJ, Burgel PR, Tomaszewski EL, Mullerova H, Reddel HK; NOVELTY study investigators. Frequent productive cough: Symptom burden and future exacerbation risk among patients with asthma and/or COPD in the NOVELTY study. Respir Med. 2022 Aug-Sep;200:106921. doi: 10.1016/j.rmed.2022.106921. Epub 2022 Jun 20. PMID 35820227
- [Derived] Reddel HK, Vestbo J, Agusti A, Anderson GP, Bansal AT, Beasley R, Bel EH, Janson C, Make B, Pavord ID, Price D, Rapsomaniki E, Karlsson N, Finch DK, Nuevo J, de Giorgio-Miller A, Alacqua M, Hughes R, Mullerova H, Gerhardsson de Verdier M; NOVELTY study investigators. Heterogeneity within and between physician-diagnosed asthma and/or COPD: NOVELTY cohort. Eur Respir J. 2021 Sep 23;58(3):2003927. doi: 10.1183/13993003.03927-2020. Print 2021 Sep. PMID 33632799
- [Derived] Karlsson N, Atkinson MJ, Mullerova H, Alacqua M, Keen C, Hughes R, Janson C, Make B, Price D, Reddel HK; NOVELTY study investigators. Validation of a diagnosis-agnostic symptom questionnaire for asthma and/or COPD. ERJ Open Res. 2021 Feb 1;7(1):00828-2020. doi: 10.1183/23120541.00828-2020. eCollection 2021 Jan. PMID 33569501
- [Derived] Reddel HK, Gerhardsson de Verdier M, Agusti A, Anderson G, Beasley R, Bel EH, Janson C, Make B, Martin RJ, Pavord I, Price D, Keen C, Gardev A, Rennard S, Svereus A, Bansal AT, Brannman L, Karlsson N, Nuevo J, Nyberg F, Young SS, Vestbo J. Prospective observational study in patients with obstructive lung disease: NOVELTY design. ERJ Open Res. 2019 Feb 1;5(1):00036-2018. doi: 10.1183/23120541.00036-2018. eCollection 2019 Feb. PMID 30723727
- See also: NOVELTY_protocol_v1_with_amendment_history_REDACTED — https://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3871&filename=NOVELTY_protocol_v1_with_amendment_history_REDACTED.PDF
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D2287R00103&attachmentIdentifier=14e89c23-6c81-4774-b7eb-21d01690f535&fileName=D2287R00103_Year_5_Synopsis_v1_1Oct2024_Clean_Redacted.pdf&versionIdentifier=